CLINICAL TRIAL: NCT05772026
Title: Serum Biomarkers for Postoperative Delirium Based on Plasma Proteomic Analysis of Elder Patients Undergoing Cardiac Surgery
Brief Title: Plasma Proteomics in Patients With Postoperative Delirium
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XuzhouCH2023
Record Dates: First submitted 2023-02-18; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD group: According to the occurrence of postoperative delirium, the patients were divided into POD group and non-POD group
- non-POD group: According to the occurrence of postoperative delirium, the patients were divided into POD group and non-POD group

SUMMARY:
Patients undergoing cardiac surgery were recruited. Baseline characteristics of all subjects were collected. The 3-minute Delirium diagnostic Scale (3D-CAM) was used to screen the POD group and non-POD group from the recruited subjects during the first 7 days after surgery. Peripheral blood samples were collected 1 day before surgery and 2 day after surgery. . Plasma was isolated from peripheral blood for subsequent proteomic analysis.

DETAILED DESCRIPTION:
Patients undergoing noncardiac surgery were recruited. Baseline characteristics of all subjects were collected. The 3-minute Delirium diagnostic Scale (3D-CAM) was used to screen the POD group and non-POD group from the recruited subjects during the first 7 days after surgery. Peripheral blood samples were collected 1 day before surgery and 2 day after surgery. Plasma was isolated from peripheral blood for subsequent proteomic analysis. To study the characteristics of proteins on a large scale, including protein expression levels, post-translational modifications, protein-protein interactions, etc., so as to obtain a comprehensive understanding of disease occurrence, cell metabolism and other processes at the protein level. Assessment of imbalanced protein expression in peripheral blood using protein profiling may allow us to better understand the pathological changes occurring at the molecular level of POD. Early detection of patients at high risk of POD can optimize perioperative management and promote rapid postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old, regardless of gender.
* The patient had clear consciousness and no cognitive impairment, and could cooperate with the investigation and follow-up.
* The ASA classification is I-Ⅲ.

Exclusion Criteria:

* severe neurological or psychiatric disorders.
* drug and alcohol abuse.
* Patients with cognitive impairment caused by various reasons such as neuropsychiatric symptoms.
* Exclusion criteria included incomplete medical records and failure to complete the postoperative follow-up.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients undergoing cardiac Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Differences of Quantitative Proteomics between POD and non-POD | 1 day before surgery
  Plasma was isolated from peripheral blood for subsequent proteomic analysis. Investigators study the characteristics of proteins at a large-scale level.
Differences of Quantitative Proteomics between POD and non-POD after surgery | 2 day after surgery
  Plasma was isolated from peripheral blood for subsequent proteomic analysis. Investigators study the characteristics of proteins at a large-scale level.

CONTACTS AND LOCATIONS:
Overall Officials: Yangzi Zhu, Doctor, Study Director — Xuzhou Central Hospital; Liwei Wang, Doctor, Principal Investigator — Xuzhou Central Hospital

IPD SHARING:
Plan to Share IPD: No